CLINICAL TRIAL: NCT06961474
Title: Effectiveness of Treatments for Cirrhosis With Varicose Veins：A Prospective Observational Study
Brief Title: Effectiveness of Treatments for Cirrhosis With Varicose Veins
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2022-109
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Varices Bleeding; Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic treatment group
  Interventions: Procedure: Endoscopic treatment
- Non-endoscopic treatment group

INTERVENTIONS:
Procedure: Endoscopic treatment — The endoscopic treatment methods for patients with esophageal variceal rupture bleeding usually include variceal ligation and injection of tissue adhesive.
  Groups: Endoscopic treatment group

SUMMARY:
Liver cirrhosis is the fifth leading cause of death among adults, characterized by diffuse fibrous tissue proliferation and the formation of regenerative nodules and false lobules on the basis of widespread hepatocyte necrosis, leading to severe complications such as portal hypertension and liver failure. Cirrhosis is categorized into compensated and decompensated stages based on the presence or absence of clinical events such as ascites, variceal rupture bleeding, and hepatic encephalopathy. Patients with decompensated cirrhosis have a significantly shorter median survival time compared to those in the compensated stage. Esophagogastric variceal hemorrhage is a common life-threatening complication in patients with portal hypertension due to cirrhosis, with high incidence rates and mortality. Current preventive and therapeutic approaches for variceal bleeding include pharmacological therapy, endoscopic treatment, transjugular intrahepatic portosystemic shunt (TIPS), and surgical interventions. However, mortality remains high, and each treatment modality has its own limitations and controversies.

This study aims to prospectively investigate the clinical characteristics of portal hypertension caused by various etiologies (e.g., hepatitis B, autoimmune diseases, schistosomiasis) and to compare the efficacy and safety of endoscopic and interventional treatments for varices, providing evidence-based medical support for clinical diagnosis and treatment. The study includes patients admitted for portal hypertension-related esophagogastric varices from February 2022 to December 2024, excluding those under 18 years of age, without varices, or with incomplete medical records. Baseline data, including demographic features, medical history, laboratory tests, imaging examinations, and Child-Pugh classification, will be collected. Follow-up assessments will be conducted at 1, 2, 6, and 12 months post-treatment to monitor adverse events (e.g., rebleeding, hepatic encephalopathy, ascites) and survival status. The primary endpoint is the rebleeding rate within one year, while secondary endpoints include mortality and the incidence of portal hypertension-related complications.

The sample size is estimated at 1,900 patients, with 1,500 in the endoscopic treatment group and 400 in the non-endoscopic treatment group. Statistical analysis will be performed using SPSS 24.0 and R software, with continuous data analyzed using t-tests or rank-sum tests and categorical data analyzed using chi-square tests or Fisher's exact test. The study has been approved by the ethics committee, and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

① Age greater than 18 years, with no gender restriction.

② Patients admitted for portal hypertension-related esophageal and gastric varices from February 2022 to December 2024.

Exclusion Criteria:

* Age < 18 years ② Absence of esophageal or gastric varices ③ Incomplete medical history records

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted for portal hypertension-related esophageal and gastric varices from February 2022 to December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rebleeding within one year | 1 year

SECONDARY OUTCOMES:
Mortality within 1 year and the occurrence of portal hypertension-related complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Ph.D., Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China